CLINICAL TRIAL: NCT04959240
Title: Expanded Access to Velmanase Alfa
Status: Available | Type: Expanded Access
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: Velmanase alfa-EAP
Record Dates: First submitted 2021-07-01; First posted 2021-07-13 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Alpha-Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Velmanase Alfa
  Other Names: Lamzede; Lamazym; rhLAMAN; recombinant human alpha-mannosidase

SUMMARY:
Individual patient expanded access requests may be considered for patients who have no other treatment options.

DETAILED DESCRIPTION:
Expanded access may provide access for treatment prior to approval by the local regulatory agency.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult